CLINICAL TRIAL: NCT00512746
Title: A Randomised Controlled Trial of Surveillance for the Early Detection of Lung Cancer in an at Risk Group [Lung-SEARCH Trial]
Brief Title: Screening for Lung Cancer in Current or Past Smokers With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CDR0000558413; CRUK-BRD/06/10; EU-20738; ISRCTN80745975
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Lung Cancer; Precancerous Condition
Keywords: small cell lung cancer; non-small cell lung cancer; precancerous condition
MeSH Terms: conditions — Lung Neoplasms; Precancerous Conditions; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Cytological Techniques; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surveillance (Other): Screened arm
  Interventions: Other: cytology and cytometry specimen collection procedure; Other: Chest x ray; Procedure: Autofluorescence bronchoscopy; Procedure: CT scan
- Control (Active Comparator): Control arm
  Interventions: Other: Chest x ray

INTERVENTIONS:
Other: cytology and cytometry specimen collection procedure — Samples tested and further interventions added if positive
  Arms: Surveillance
Other: Chest x ray — Patients not diagnosed with lung cancer during the course of the study, will be offered an exit chest x-ray after 5 years or sooner if they withdraw from the trial before 5 years. This could help identify a lung cancer that may not have been associated with symptoms earlier.
Procedure: Autofluorescence bronchoscopy — The bronchial tree will be inspected first under white light and then under blue light. All areas that appear abnormal will initially be documented and only sampled when the bronchoscopic examination has been completed.
  Other Names: AFB
  Arms: Surveillance
Procedure: CT scan — All patients with abnormal sputum cytology and/or cytometry will undergo low dose spiral CT without contrast.
  Arms: Surveillance

SUMMARY:
RATIONALE: Screening tests or exams may help doctors find lung cancer sooner, when it may be easier to treat.

PURPOSE: This randomized clinical trial is studying screening tests or exams to see how well they work compared to usual care in finding early stage lung cancer in current or past smokers with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To show that the proportion of lung cancer diagnosed at stage I or II is significantly greater in the surveillance arm than in the control arm.

Secondary

* Establish whether sputum cytology and/or cytometry can be employed to stratify patients with chronic obstructive pulmonary disease (COPD) according to their risk of developing incidence lung cancer.
* Identify patients with pre-invasive lesions in their airways and examine the risk of developing lung cancer in patients harboring these lesions.
* Provide an opportunity to archive blood samples from patients under surveillance to enable the identification of markers of disease progression.
* Examine the compliance of regular screening among patients in this high-risk group.
* Determine the proportion of patients in which it is not possible to provide a sputum screening result.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to recruiting site, age, gender, smoking history (current vs ex-smoker) and severity of chronic obstructive pulmonary disease (COPD) (mild vs moderate). Patients are randomized to 1 of 2 arms.

* Control arm: Patients are managed according to the usual practice of their hospital or general practice for their COPD treatment. They undergo no particular investigations except those that may arise due to a change in their clinical condition. Those patients who are not diagnosed with lung cancer during the course of the study are offered a chest x-ray after 5 years of follow-up.
* Surveillance arm: Patients undergo surveillance for 5 years. A sputum sample is collected for cytology and cytometry. If the sputum sample is normal the patient is asked to provide a sputum sample annually. If the sputum sample is abnormal the patient undergoes an annual spiral CT scan followed by autofluorescence bronchoscopy. At bronchoscopy, the following samples are taken: bronchial washings, bronchial brushings, and bronchial biopsies. Bronchoscopy is repeated every 4-12 months depending upon the histology results. If an invasive lesion is found, the patient is referred for treatment via the normal hospital systems. Any remaining sputum sample is stored frozen as part of the tissue bank associated with this trial.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Meets 1 of the following criteria:

  * Current smoker, defined as ≥ a 20 pack year smoking history and/or 20 year duration of smoking
  * Ex-smoker who has quit smoking within the past 8 years AND has ≥ a 20 pack year smoking history and/or 20 year duration of smoking
* Mild to moderate chronic obstructive pulmonary disease (COPD) as defined by the GOLD criteria

  * Mild COPD: FEV_1/forced vital capacity (FVC) < 70%; FEV_1 ≥ 80% of predicted*
  * Moderate COPD: FEV_1/FVC < 70%; FEV_1 50-80% of predicted* NOTE: *Spirometric values will be obtained post bronchodilator according to the recommendations in the GOLD criteria

Exclusion criteria:

* Inadequate lung function (FEV_1 < 50% of predicted after bronchodilator)

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Life expectancy must be at least 5 years

Exclusion criteria:

* History of malignant disease within the past 5 years except non-melanomatous skin cancers
* Other serious co-morbidity
* Evidence of severe or uncontrolled systemic diseases that, in the view of the investigator, makes it undesirable for the patient to participate in this trial
* Any disorder making reliable informed consent impossible
* Unlikely to co-operate with a 5 year follow-up

PRIOR CONCURRENT THERAPY:

* Patients may receive all concurrent therapy deemed to provide adequate care as decided by their medical doctors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1569 (Actual)
Dates: Start 2007-08; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Proportion of lung cancer that is diagnosed as stage I or II | 5 years
  In the control arm, it is expected that only 15% of cancers will be detected early. In the surveillance arm, we expect that at the time of the first screen, the detection rate of prevalence cancers will be about 3%, from data reported in CT screening studies

SECONDARY OUTCOMES:
Uptake of screening (the proportion of patients in the surveillance arm who undergo annual screening, among those invited to attend) | 5 Years
Proportion of patients in the surveillance arm who have abnormal sputum cytology | 5 Years
Proportion of patients in the surveillance arm who have abnormal sputum cytometry | 5 Years
Death from lung cancer | Up to 15 years
Proportion of failed sputum samples (i.e., where it is not possible to obtain adequate sputum samples) | 5 Years
Prevalence of pre-invasive disease in patients in the surveillance arm with abnormal cytometry | 5 Years
Number of patients in the surveillance arm with pre-invasive lesions who develop lung cancer locally and at remote sites within the lung | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G. Spiro, Study Chair — University College London Hospitals
Locations (10):
- United Kingdom (10):
  - Papworth Hospital, Cambridge, England
  - Walsgrave Hospital, Coventry, England
  - Leeds General Infirmary, Leeds, England
  - University Hospitals of Leicester NHS Trust, Leicester, England
  - Chelsea Westminster Hospital, London, England
  - Royal Brompton Hospital, London, England
  - University College Hospital - London, London, England
  - Wythenshawe Hospital, Manchester, England
  - Sunderland Royal Hospital, Sunderland, England
  - Respiratory Research Office Belfast City Hospital, Belfast, Northern Ireland

REFERENCES:
- [Derived] Spiro SG, Hackshaw A; LungSEARCH Collaborative Group. Research in progress--LungSEARCH: a randomised controlled trial of surveillance for the early detection of lung cancer in a high-risk group. Thorax. 2016 Jan;71(1):91-3. doi: 10.1136/thoraxjnl-2015-207433. Epub 2015 Jul 2. PMID 26138736